CLINICAL TRIAL: NCT07101783
Title: Investigation of Pharmacokinetic Properties of Single Doses of NNC0662-0419 in Japanese, Chinese and Non-Asian Participants Living With Overweight or Obesity
Brief Title: A Research Study on How a Dose of NNC0662-0419 Works in Japanese, Chinese and Non-Asian Participants Living With Overweight or Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9662-8159; U1111-1315-2937 (Other: World Health Organization (WHO))
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- NNC0662-0419 (Dose 1) (Experimental): Participants will receive a single dose (SD) of NNC0662-0419 subcutaneously.
  Interventions: Drug: NNC0662-0419
- NNC0662-0419 (Dose 2) (Experimental): Participants will receive a SD of NNC0662-0419 subcutaneously.
  Interventions: Drug: NNC0662-0419
- NNC0662-0419 (Dose 3) (Experimental): Participants will receive a SD of NNC0662-0419 subcutaneously.
  Interventions: Drug: NNC0662-0419

INTERVENTIONS:
Drug: NNC0662-0419 — Participants will receive NNC0662-0419 subcutaneously.

SUMMARY:
The study is testing the new medicine NNC0662-0419 in people living with overweight or obesity. The purpose of the study is to look into the amount of the new medicine NNC0662-0419 in participants blood after one dose. And also look into how safe and how well the study medicine is tolerated in people living with overweight or obesity. NNC0662-0419 is a new medicine which cannot be prescribed by doctors. NNC0662-0419 is currently being tested in humans and the dose participants will receive has been found safe and tolerable. Participants will get a single dose of NNC0662-0419 given by study staff as a single injection under participants skin. Like all medicines, the study medicine may have side effects. The study will last up to 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female (sex at birth) Japanese, Chinese or non-Asian participants (all self-reported).

  * For Japanese participants: both parents of Japanese descent.
  * For Chinese participants: both parents of Chinese descent.
  * For non-Asian participants: both parents of non-Asian descent (non-Asian is defined as of countries outside of Asia).
* Age 18-55 years (both inclusive) at the time of signing the informed consent.
* Body mass index (BMI) between 24.0 and 34.9 kilogram per square meter (kg/m^2) (both inclusive) at screening. Overweight should be due to excess adipose tissue, as judged by the investigator.
* Considered eligible based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Exclusion Criteria:

* Known a* or suspected hypersensitivity to study intervention(s) or related products.
* Any disorder, unwillingness or inability which in the investigator's opinion, might jeopardise the participant's safety or compliance with the protocol.
* 2nd or 3rd degree atrioventricular-block, prolongation of the QRS complex over 120 millisecond (msec), or of the corrected QT interval by Fridericia (QTcF) calculation over 450 msec (females) or 430 msec (males), or any other clinically significant abnormal electrocardiogram (ECG) results as judged by the investigator, at screening.
* Glycated haemoglobin (HbA1c) greater than or equal to >= 6.5percent (%) (48 millimoles per liter [mmol/mol]) at screening.
* Calcitonin >= 50 nanogram per liter (ng/L) at screening. a* - As declared by the participant or reported in the medical records.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
AUC; The area under the NNC0662-0419 plasma concentration-time curve | From pre-dose on Day 1 until completion of the end of study visit (Day 29)
  Measured in hours*nanomoles per liter (h*nmol/L).

SECONDARY OUTCOMES:
Cmax; The maximum plasma concentration of NNC0662-0419 | From pre-dose on Day 1 until completion of the end of study visit (Day 29)
  Measured in nanomoles per liter (nmol/L).
Number of treatment-emergent adverse events (TEAEs) | From time of dosing on Day 1 until completion of the end of study visit (Day 29)
  Measured as number of events.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Altasciences Clinical LA, Inc., Cypress, California, United States

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com.
URL: http://novonordisk-trials.com